CLINICAL TRIAL: NCT02591381
Title: A Randomized Study of Transcorporal Versus Standard Artificial Urinary Sphincter Placement
Brief Title: Transcorporal Versus Standard Artificial Urinary Sphincter Placement
Acronym: TC vs ST AUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was started but closed prior to completion because we could not meet enrollment numbers
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Minnesota (Other); Baylor College of Medicine (Other); University of Iowa (Other); University of Kansas (Other); Central Ohio Urology Group (Other); Loyola University Chicago (Other); Lahey Clinic (Other); University of Washington (Other); New York University (Other); University of California, San Diego (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Benjamin Breyer, MD, Chief of Urology, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K12DK083021-AUS; K12DK083021 (NIH)
Record Dates: First submitted 2015-10-20; First posted 2015-10-29 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Urinary Stress Incontinence
Keywords: urinary stress incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STANDARD AUS Placement (Experimental): Standard placement of an artificial urinary sphincter involves a small incision made in the patient's perineum or scrotum and a fluid-filled cuff is placed around the bulbar urethra (the portion of the urethra between the bladder neck and penis). Connected to the cuff with tubing, is a balloon filled with fluid that is placed behind the pubic bone or in the space between the peritoneum and abdominal muscles. A control pump is placed in the scrotum and allows the device to cycle, thus either exerting pressure to close off the urethra or releasing pressure to allow the urethra to open and the patient to void.
  Interventions: Procedure: Artificial Urinary Sphincter Placement
- TRANSCORPORAL AUS Placement (Experimental): Transcorporal placement has been introduced as a way to reduce risk of erosion and involves tunneling the cuff through the erectile bodies. The same incision is made as for the standard approach, and then an incision is made in each corpus cavernosum (cylinders of tissue that allow for erection). This allows the cuff to be placed around both the urethra and through the lining of the corporal bodies, increasing the bulk of tissue behind the urethra to protect it from erosion.
  Interventions: Procedure: Artificial Urinary Sphincter Placement

INTERVENTIONS:
Procedure: Artificial Urinary Sphincter Placement — The AUS is the gold standard for treatment of severe stress urinary incontinence, particularly in patients following surgical resection of the prostate for prostate cancer. AUSs are small devices that prevent urinary flow via compression of the urethra, thus mimicking the native urinary sphincter.

SUMMARY:
The investigators propose a randomized non-blinded comparison of standard vs. transcorporal approach for placement of an artificial urinary sphincter in male patients with stress urinary incontinence after radiation and radical prostatectomy for prostate cancer. In the United States, the artificial urinary sphincter (AUS), manufactured by American Medical Systems, is the gold standard surgical treatment for stress urinary incontinence (SUI) in men. The cuff, which is the portion of the device that encircles and occludes the urethra, is typically placed directly around the urethra (i.e., "standard" placement). The cuff can erode into the urethra. Transcorporal placement has been introduced as a method to reduce the risk of erosion. Transcorporal placement involves tunneling the cuff through the erectile bodies so as to protect the dorsal aspect of the urethra. This approach has never been compared to standard placement in a randomized fashion. In the randomized trial, no additional procedures beyond the normal care protocol will be required of the patients. The investigators will conduct the study through an established, IRB-approved multi-institutional network of surgeons. Success will be assessed via objective and subjective methods; complications will be tallied in a standardized fashion. Outcomes will be measured at two years.

DETAILED DESCRIPTION:
Procedure/ Methods:

Patients will be identified in the urology clinic upon their standard of care visit for AUS placement. The procedures that determine whether a patient is a surgical candidate are as follows:

* Incontinence Impact Questionnaire Short Form (IIQ-7) and Urinary Incontinence Symptoms index (ISI) standardized questionnaires
* Physical examination
* Review of medical history that would preclude surgery
* Cystoscopy to evaluate and rule out stricture
* Uroflow/Post void residual to ensure adequate bladder capacity

Pre surgery work up includes:

* Urine analysis and if indicated urine culture and treatment of urinary tract infection
* Flow, post-void residual if possible
* Cystoscopy to rule out bladder neck contracture or urethral stricture
* History and physical examination
* Treatment of men with 2 days of chlorhexidine wash to the perineum
* Incontinence sexual function questionaires
* Aminogllycoside and other abx prior to surgery
* 24 hour pad weight

Post-surgery follow up:

* Routine removal of catheter within 5 days post-op
* Treatment of antibiotics post-operatively to be limited to 1 week
* Activation of AUS at 4-8 weeks post-op
* Incontinence sexual function questionnaires
* 24 hour pad weight

Routine follow ups will be conducted at 2 weeks, 6 weeks, 3 months, 6 months post-operatively, and yearly thereafter (SOC). Patient characteristics that will be collected include:

* etiology of the incontinence.
* pre-operative pad usage
* prior anti-incontinence procedures
* adjuvant therapy for prostate cancer such as radiotherapy, or other history of pelvic radiation
* post-operative urodynamic studies
* cystoscopy findings

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing an AUS procedure would potentially be candidates for the study

Exclusion Criteria: There are several situations in which either a TC or ST procedure would be specifically indicated, and it would be unethical to randomize these patients to the other procedure.

* No men without erectile dysfunction
* No use of injectable agents into the corporal body
* No prior urethral surgery (Prior surgery defined as; urethroplasty, urethral sling, prior AUS placement or explantation, recto-urethral fistula closure)
* No current penile prosthesis
* No concomitant placement of penile prosthesis at the time of AUS placement
* Males under the age of 18, as well as females, are also excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Revision or removal surgery for AUS cuff problems other than mechanical failure: these include cuff erosion, impending erosion (discretion of surgeon), persistent retention due to small cuff, urethral atrophy | Through study completion, an average of up to 1 year

SECONDARY OUTCOMES:
Rate of post-operative urinary retention | Up to 2-4 weeks
  Urinary retention defined as urinary catheter placement for more than 5 days post-op.
Change in 24 hour pad test at 3 months post-op compared to pre-op | 3 months post op
Erectile function as measured pre and post AUS placement via the Sexual Health Inventory for Men (SHIM) | 3 month post op, 12 month post op
  Sexual health is an important part of an individual's overall physical and emotional well being. This questionnaire is designed to help identify if the patient may be experiencing erectile dysfunction.
Incontinence impact as measured by the Incontinence Symptom Index (ISI) | 3 month post op, 12 month post op
  This brief questionnaire is designed to assess the severity of the patient's urinary incontinence
Quality of Life impact as measured by the Incontinence Impact Questionnaire--Short Form (IIQ) | 3 month post op, 12 month post op
  Some people find that accidental urine loss may affect their activities, relationships, and feelings. The questions in this assessment refer to areas in the subjects life that may have been influenced or changed by incontinent symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: benjamin n breyer, MD, MAS, FAC, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Haab F, Trockman BA, Zimmern PE, Leach GE. Quality of life and continence assessment of the artificial urinary sphincter in men with minimum 3.5 years of followup. J Urol. 1997 Aug;158(2):435-9. PMID 9224318
- [Background] Dalkin BL, Wessells H, Cui H. A national survey of urinary and health related quality of life outcomes in men with an artificial urinary sphincter for post-radical prostatectomy incontinence. J Urol. 2003 Jan;169(1):237-9. doi: 10.1016/S0022-5347(05)64076-1. PMID 12478144
- [Background] Guralnick ML, Miller E, Toh KL, Webster GD. Transcorporal artificial urinary sphincter cuff placement in cases requiring revision for erosion and urethral atrophy. J Urol. 2002 May;167(5):2075-8; discussion 2079. PMID 11956443
- [Background] Aaronson DS, Elliott SP, McAninch JW. Transcorporal artificial urinary sphincter placement for incontinence in high-risk patients after treatment of prostate cancer. Urology. 2008 Oct;72(4):825-7. doi: 10.1016/j.urology.2008.06.065. Epub 2008 Aug 26. PMID 18752838